CLINICAL TRIAL: NCT05580107
Title: Open-label Phase Ib Study of Preoperative Treatment With the KLK Inhibitor MDPK67b in Patients With Untreated Prostate Cancer
Brief Title: MDPK67b in Patients With Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Med Discovery SA (Industry)
Collaborators: Camara and Partners Sàrl (Unknown); Soladis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MDPK67b-2002
Record Dates: First submitted 2022-07-07; First posted 2022-10-14 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy; Gleason score 7 or higher
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose finding (24 and 48 mg) based on dose limiting toxicity (DLT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose (Experimental): Five patients will be included into the 24 mg dose level. In case of dose limiting toxicity (DLT) in at least one patient, 5 additional patients will be enrolled in the 24 mg dose level.
  If the treatment is well tolerated, i.e. no DLT is encountered, the dose of MDPK67b is escalated to 48 mg on a second cohort of 5 patients. In case of DLT in at least one patient at the 48 mg dose level, the 24 mg dose level of MDPK67b is expanded from 5 to 10 patients, or declared the maximum tolerated dose (MTD) if already expanded to 10 patients.
  Interventions: Drug: MDPK67b

INTERVENTIONS:
Drug: MDPK67b — 24 mg or 48 mg

SUMMARY:
Administration of MDPK67b to assess its Tolerability and Safety profile in prostate cancer patients, and to assess histo-pathological and molecular changes in prostate tumor tissue samples.

ELIGIBILITY:
Subject screening criteria

1. Patients aged 18 years or older.
2. Patients who have untreated suspected PCa or PCa under active surveillance (AS) with progression/upgrading.
3. Patients who signed a written screening phase ICF.

Subject non-screening criteria

1. Patients who have an uncontrolled disease that would unduly increase the risk of toxicity or limit compliance with study requirements in the opinion of the Investigator; including but not limited to: ongoing or active symptomatic infection, uncontrolled diabetes mellitus, diseases of the coagulation system, unstable or uncompensated cardiac, hepatic, renal, respiratory, or psychiatric disease.
2. Patients who required a significant change in their concomitant medications during the week prior to screening visit, or who will likely need to have a change in their concomitant medications during the study. This includes any medication other than those required for PCa diagnosis or for RPE.
3. Patients who have received prior radiotherapy to the prostate.
4. Patients who have had prior exposure to MDPK67b.
5. Patients who have participated in another clinical trial within 3 months prior to screening visit, except if in the opinion of the investigator the type of trial does not interfere in any way with the present trial (eg. non-interventional observational trial). In case of doubt, the sponsor's prior approval must be obtained and the decision to include such a patient will be documented in detail.

Non-screening criteria are exclusion criteria for the screening phase.

For the patients not participating in the screening phase (ie patients with previously established PCa diagnosis), all the criteria above shall be checked prior to enrolment in the treatment phase. However, these patients do not have to sign a screening ICF (screening criterion n°3 is not applicable), and for non-screening criterion n°5, the 3-month wash-out period is prior to the inclusion visit in the treatment phase.

Subject inclusion criteria

1. Patients who still meet all the eligibility criteria checked at screening visit.
2. Patients who have untreated PCa with a Gleason score of 7 (preferably) or higher, with local disease or with metastatic disease (if metastatic, no visceral metastases, no more than five bone or lymph node metastases), and are scheduled to undergo RPE about 3 weeks later.
3. Patients with an expected minimal survival time of 12 months.
4. Patients who have an acceptable organ and marrow function as assessed at the inclusion visit and defined as follows:

   1. Absolute neutrophil count ≥ 1.5 × 109/L.
   2. Platelets ≥ 100 × 109/L.
   3. Hemoglobin ≥ 9 g/dL.
   4. Total bilirubin ≤ 1.5 × ULN, unless the patient has known Gilbert's syndrome.
   5. Aspartate amino transferase (AST) and alanine amino transferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN in presence of liver metastasis.
   6. Serum creatinine ≤ 2.0 × ULN, or GFR ≥ 30 mL/min by Cockcroft-Gault.
   7. INR <1.5, aPTT < 60 s
5. Patients with an ECOG performance status ≤ 1.
6. Patients who agree to refrain to donate sperm for the duration of the study.
7. Patients who signed a written treatment phase ICF.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Tolerability and Safety | Day 1
  Number of subjects with changes in blood pressure
Tolerability and Safety | Day 8
  Number of subjects with changes in blood pressure
Tolerability and Safety | Day 15
  Number of subjects with changes in blood pressure
Tolerability and Safety | Day 20-25
  Number of subjects with changes in blood pressure
Tolerability and Safety | Day 1
  Body temperature
Tolerability and Safety | Day 8
  Number of subjects with changes in body temperature
Tolerability and Safety | Day 15
  Number of subjects with changes in body temperature
Tolerability and Safety | Day 20-25
  Number of subjects with changes in body temperature
Tolerability and Safety | Day 1
  Number of subjects with changes in respiration rate
Tolerability and Safety | Day 8
  Number of subjects with changes in respiration rate
Tolerability and Safety | Day 15
  Number of subjects with changes in respiration rate
Tolerability and Safety | Day 20-25
  Number of subjects with changes in respiration rate
Tolerability and Safety | Day 1
  Number of subjects with changes in weight
Tolerability and Safety | Day 8
  Number of subjects with changes in weight
Tolerability and Safety | Day 15
  Number of subjects with changes in weight
Tolerability and Safety | Day 20-25
  Number of subjects with changes in weight
Tolerability and Safety | Day 1
  Number of subjects with changes in QTc on ECG
Tolerability and Safety | Day 8
  Number of subjects with changes in QTc on ECG
Tolerability and Safety | Day 15
  Number of subjects with changes in QTc on ECG
Tolerability and Safety | Day 20-25
  Number of subjects with changes in QTc on ECG
Tolerability and Safety | Day 1
  Number of subjects with changes in heart rate on ECG
Tolerability and Safety | Day 8
  Number of subjects with changes in heart rate on ECG
Tolerability and Safety | Day 15
  Number of subjects with changes in heart rate on ECG
Tolerability and Safety | Day 20-25
  Number of subjects with changes in heart rate on ECG
Tolerability and Safety | Day 8
  Number of subjects with changes in hematology safety parameters: haemoglobin, haematocrit, RBC, MCH, MCV, WBC differential count (absolute and relative count), platelet count, INR, aPTT, Thrombin time and fibrinogen
Tolerability and Safety | Day 15
  Number of subjects with changes in hematology safety parameters: haemoglobin, haematocrit, RBC, MCH, MCV, WBC differential count (absolute and relative count), platelet count, INR, aPTT, Thrombin time and fibrinogen
Tolerability and Safety | Day 20-25
  Number of subjects with changes in hematology safety parameters: haemoglobin, haematocrit, RBC, MCH, MCV, WBC differential count (absolute and relative count), platelet count, INR, aPTT, Thrombin time and fibrinogen
Tolerability and Safety | Day 8
  Number of subjects with changes in blood chemistry safety parameters: fasting glucose, total protein, creatinine, urea, sodium, potassium, calcium, uric acid, AST, ALT, CPK, AlkP, LDH, total bilirubin, PSA
Tolerability and Safety | Day 15
  Number of subjects with changes in blood chemistry safety parameters: fasting glucose, total protein, creatinine, urea, sodium, potassium, calcium, uric acid, AST, ALT, CPK, AlkP, LDH, total bilirubin, PSA
Tolerability and Safety | Day 20-25
  Number of subjects with changes in blood chemistry safety parameters: fasting glucose, total protein, creatinine, urea, sodium, potassium, calcium, uric acid, AST, ALT, CPK, AlkP, LDH, total bilirubin, PSA
Tolerability and Safety | Day 8
  Number of subjects with changes in urine safety parameters: pH, ketones, protein, glucose, blood, leukocytes, urobilinogen, bilirubin
Tolerability and Safety | Day 15
  Number of subjects with changes in urine safety parameters: pH, ketones, protein, glucose, blood, leukocytes, urobilinogen, bilirubin
Tolerability and Safety | Day 20-25
  Number of subjects with changes in urine safety parameters: pH, ketones, protein, glucose, blood, leukocytes, urobilinogen, bilirubin
Tolerability and Safety | Day 1
  Number of subjects with changes in physical examination
Tolerability and Safety | Day 8
  Number of subjects with changes in physical examination
Tolerability and Safety | Day 15
  Number of subjects with changes in physical examination
Tolerability and Safety | Day 20-25
  Number of subjects with changes in physical examination
Tolerability and Safety | Day 1
  Adverse events
Tolerability and Safety | Day 8
  Adverse events
Tolerability and Safety | Day 15
  Adverse events
Tolerability and Safety | Day 20-25
  Adverse events
Tolerability and Safety | Day 1
  Local tolerance using the 5-point Draize scale (0: no irritation to 5: Frank vein thrombosis in addition to grade 4 signs and symptoms)
Tolerability and Safety | Day 8
  Local tolerance using the 5-point Draize scale (0: no irritation to 5: Frank vein thrombosis in addition to grade 4 signs and symptoms)
Tolerability and Safety | Day 15
  Local tolerance using the 5-point Draize scale (0: no irritation to 5: Frank vein thrombosis in addition to grade 4 signs and symptoms)

SECONDARY OUTCOMES:
Histo-pathological and molecular changes in prostate tumor tissue samples | Screening (Diagnostic biopsy)
  Androgen receptor expression
Histo-pathological and molecular changes in prostate tumor tissue samples | Day 16/17 (Radical prostatectomy sample)
  Androgen receptor expression
Histo-pathological and molecular changes in prostate tumor tissue samples | Screening (Diagnostic biopsy)
  Extent of proliferation using Ki67
Histo-pathological and molecular changes in prostate tumor tissue samples | Day 16/17 (Radical prostatectomy sample)
  Extent of proliferation using Ki67
Histo-pathological and molecular changes in prostate tumor tissue samples | Screening (Diagnostic biopsy)
  Extent of inflammation using leukocyte markers
Histo-pathological and molecular changes in prostate tumor tissue samples | Day 16/17 (Radical prostatectomy sample)
  Extent of inflammation using leukocyte markers
Histo-pathological and molecular changes in prostate tumor tissue samples | Screening (Diagnostic biopsy)
  Expression of KLK2, KLK4, and KLK14 using immunohistochemistry
Histo-pathological and molecular changes in prostate tumor tissue samples | Day 16/17 (Radical prostatectomy sample)
  Expression of KLK2, KLK4, and KLK14 using immunohistochemistry
Histo-pathological and molecular changes in prostate tumor tissue samples | Screening (Diagnostic biopsy)
  Treatment induced change in RNA transcriptome assessed by RNA sequencing
Histo-pathological and molecular changes in prostate tumor tissue samples | Day 16/17 (Radical prostatectomy sample)
  Treatment induced change in RNA transcriptome assessed by RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eberli, Prof., Principal Investigator — Klinik für Urologie, UniversitätSpital Zürich (USZ)
Locations (1):
- Klinik für Urologie, UniversitätSpital Zürich (USZ), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No